CLINICAL TRIAL: NCT04720586
Title: Lower Eyelid Retractors Plication , Transcutaneous Blepharoplasty and Wedge Resection for Treatment of Lower Eyelid Involutional Entropion and Dermatochalasis
Brief Title: Surgical Treatment of Lower Eyelid Involutional Entropion and Dermatochalasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hamaky9
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Eyelid Diseases
Keywords: entropion; blepharoplasty
MeSH Terms: conditions — Eyelid Diseases; Entropion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- triple procedure (Experimental): lower eyelid retractors plication , transcutaneous blepharoplasty and wedge resection
  Interventions: Procedure: lower eyelid blepharoplasty , retractor plication and wedge resection; Procedure: lower eyelid blepharoplasty and retractor plication
- combined procedure (Active Comparator): lower eyelid retractors plication and transcutaneous blepharoplasty
  Interventions: Procedure: lower eyelid blepharoplasty , retractor plication and wedge resection; Procedure: lower eyelid blepharoplasty and retractor plication

INTERVENTIONS:
Procedure: lower eyelid blepharoplasty , retractor plication and wedge resection — combined lower eyelid blepharoplasty , retractor plication and wedge resection
Procedure: lower eyelid blepharoplasty and retractor plication — combined lower eyelid blepharoplasty and retractor plication procedures

SUMMARY:
lower eyelid involutional entropion and dermatochalasis are common associated problems. combined approaches give good results.

DETAILED DESCRIPTION:
traditional lower eyelid transcutaneous blepharoplasty ; subciliary incision followed by proper dissection then lower eyelid retractors plication after orbital fat removal . pentagon wedge resection of lateral lower eyelid is done

ELIGIBILITY:
Inclusion Criteria:

1. Lower eyelid involutional entropion
2. dermatochalasis

Exclusion Criteria:

1. Other eyelid disease,
2. Other causes of entropion
3. Previous eyelid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale | 12 months
  calculate scale score (1-5); score 1 is exceptional improvement , score 5 is worsened patient

CONTACTS AND LOCATIONS:
Overall Officials: Tarek R Elahamky, MD, Principal Investigator — Benaha university faculty of medicine
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates